CLINICAL TRIAL: NCT06984094
Title: A Phase 1, Randomized, Observer-blind, First-in-human Study to Describe the Safety, Reactogenicity and Immunogenicity of SCB-1022 and SCB-1033 in Healthy Older Adults Aged 60-85 Years
Brief Title: First-in-human Safety and Immunogenicity Study of SCB-1022 and SCB-1033 in Healthy Older Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-1033-001
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Syncytial Virus Vaccination; Human Metapneumovirus Vaccination; Parainfluenza Vaccination
Keywords: Respiratory Syncytial Virus vaccination; Human Matapneumovirus vaccination; Parainfluenza vaccination; healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1 (SCB-1022 dose level 1) (Experimental): 24 adults to receive dose level 1 of SCB-1022 at Day 1
  Interventions: Biological: SCB-1022
- Group 2 (SCB-1022 dose level 2) (Experimental): 24 adults to receive dose level 2 of SCB-1022 at Day 1
  Interventions: Biological: SCB-1022
- Group 3 (SCB-1033 dose level 1) (Experimental): 24 adults to receive dose level 1 of SCB-1033 at Day 1
  Interventions: Biological: SCB-1033
- Group 4 (SCB-1019T) (Active Comparator): 24 adults to receive SCB-1019T at Day 1
  Interventions: Biological: SCB-1019T
- Group 5 (SCB-1022 dose level 3) (Experimental): 24 adults to receive dose level 3 of SCB-1022 at Day 1
  Interventions: Biological: SCB-1022
- Group 6 (SCB-1033 dose level 2) (Experimental): 24 adults to receive dose level 2 of SCB-1033 at Day 1
  Interventions: Biological: SCB-1033
- Group 7 (SCB-1033 dose level 3) (Experimental): 24 adults to receive dose level 3 of SCB-1033 at Day 1
  Interventions: Biological: SCB-1033
- Group 8 (SCB-1019T) (Active Comparator): 24 adults to receive SCB-1019T at Day 1
  Interventions: Biological: SCB-1019T

INTERVENTIONS:
Biological: SCB-1019T — SCB-1019T (bivalent recombinant RSV vaccine candidate) consists of two recombinant protein subunit antigens: RSV A strain (SCB-1019T(A)) and RSV B strain (SCB-1019T(B)).
  Arms: Group 4 (SCB-1019T); Group 8 (SCB-1019T)
Biological: SCB-1022 — SCB-1022 (combination recombinant RSV-hMPV vaccine candidate) consists of three recombinant protein subunit antigens: RSV A strain (SCB-1019T(A)), RSV B strain (SCB-1019T(B)), and hMPV (SCB-1021).
  Arms: Group 1 (SCB-1022 dose level 1); Group 2 (SCB-1022 dose level 2); Group 5 (SCB-1022 dose level 3)
Biological: SCB-1033 — SCB-1033 (combination recombinant RSV-hMPV-PIV3 vaccine candidate) consists of four recombinant protein subunit antigens: RSV A strain (SCB-1019T(A)), RSV B strain (SCB-1019T(B)), hMPV (SCB-1021) and PIV3 (SCB-1020).
  Arms: Group 3 (SCB-1033 dose level 1); Group 6 (SCB-1033 dose level 2); Group 7 (SCB-1033 dose level 3)

SUMMARY:
This phase 1 study will evaluate the safety, reactogenicity, and immunogenicity of 3 different dose levels of SCB-1022 and SCB-1033 in healthy adults aged 60-85 years.

DETAILED DESCRIPTION:
The study will descriptively evaluate three dose levels of SCB-1022 and SCB-1033. The sample size for this study is not based on formal statistical hypothesis testing but is acceptable for safety and immunogenicity evaluation in a phase 1 study. The study will be overseen by a safety monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 60 to 85 years of age at the screening visit.
* Individuals willing and able to comply with study requirements, including all scheduled visits, vaccination, laboratory tests, and other study procedures.
* Individuals willing and able to give an informed consent, prior to screening.
* Healthy participants as determined by medical history, physical examination, and clinical judgment of the investigator; participants with pre-existing stable medical conditions can be included.

Please refer to Protocol for full list of Inclusion and Exclusion criteria.

Exclusion Criteria:

* Pregnancy or potential to become pregnant during the study.
* Acute disease or fever (≥38°C) at time of vaccination.
* History of Guillain-Barré Syndrome (GBS).
* Recurrent or un-controlled neurological disorders or seizures.
* Serious or unstable chronic illnesses. Please refer to Protocol for full list of Inclusion and Exclusion criteria.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and reactogenicity of SCB-1022 and SCB 1033 compared to SCB-1019T. | Within 7 days after vaccination
  Proportion of participants with local and systemic solicited AEs
To evaluate the safety and reactogenicity of SCB-1022 and SCB 1033 compared to SCB-1019T. | Within 28 days after vaccination
  Proportion of participants with unsolicited AEs
To evaluate the safety and reactogenicity of SCB-1022 and SCB 1033 compared to SCB-1019T. | Throughout the study period, from enrollment to 6 months follow up
  Proportion of participants with SAEs, AESIs, MAAEs, AEs leading to early termination from the study
To evaluate the safety and reactogenicity of SCB-1022 and SCB 1033 compared to SCB-1019T. | Screening and day 8
  Mean change and shift from baseline in hematology, biochemistry and coagulation parameters; by safety set.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Rook, MD, Principal Investigator — Fusion Clinical Research
Locations (1):
- Fusion Clinical Research, Adelaide, Southern Australia, Australia

IPD SHARING:
Plan to Share IPD: No